CLINICAL TRIAL: NCT02219477
Title: An Open-Label Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With Ribavirin in Adults With Genotype 1 and Ombitasvir/Paritaprevir/Ritonavir With Ribavirin in Adults With Genotype 4 Chronic Hepatitis C Virus Infection and Decompensated Cirrhosis (TURQUOISE-CPB)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With Ribavirin in Adults With Genotype 1 and Ombitasvir/Paritaprevir/Ritonavir With Ribavirin in Adults With Genotype 4 Chronic Hepatitis C Virus Infection and Decompensated Cirrhosis
Acronym: TURQUOISE-CPB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-227; 2014-001477-13 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Chronic Hepatitis C; Decompensated Cirrhosis; Hepatitis C Virus
Keywords: Cirrhosis; Hepatitis C; Child-Pugh B; Hepatitis C Genotype 4; Interferon-Free; Hepatitis C Genotype 1; Chronic Hepatitis C; Decompensated Cirrhosis; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — ombitasvir; paritaprevir; Ritonavir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: GT1B (Experimental): ombitasvir/paritaprevir/ritonavir 25/150/100 mg once daily (QD) + dasabuvir 250 mg twice daily (BID) + ribavirin (RBV) for 12 weeks in hepatitis C virus (HCV) genotype (GT) 1b-infected participants
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: dasabuvir; Drug: ribavirin
- Group 2: GT1 Non-B (Experimental): ombitasvir/paritaprevir/ritonavir 25/150/100 mg QD + dasabuvir 250 mg BID + RBV for 24 weeks in HCV GT1non-b (including GT1a)-infected participants
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: dasabuvir; Drug: ribavirin
- Group 3: GT4 (Experimental): ombitasvir/paritaprevir/ritonavir 25/150/100 mg QD + RBV for 24 weeks in HCV GT4-infected participants
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir — tablet; paritaprevir co-formulated with ritonavir and ombitasvir
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ritonavir also known as norvir
Drug: dasabuvir — tablet
  Other Names: ABT-333
  Arms: Group 1: GT1B; Group 2: GT1 Non-B
Drug: ribavirin — tablet

SUMMARY:
The primary objectives of this study are to assess the safety and the SVR12 rate of ombitasvir/paritaprevir/ritonavir and dasabuvir with RBV in GT1-infected participants with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. HCV GT1- or GT4-infection defined as: positive for anti-HCV Ab, HCV RNA > 1,000 IU/mL and laboratory result indicating HCV GT1 or GT4 infection at Screening.
2. Evidence of cirrhosis by prior liver biopsy, FibroScan or by radiograph (i.e., computed tomography [CT] scan or magnetic resonance imaging [MRI]).
3. Child-Pugh Score of 7 - 9, inclusive, at time of Screening.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Positive test result for Hepatitis B surface antigen (HbsAg) or anti-HIV antibodies (HIV Ab).
3. Prior or current use of any other investigational or commercially available anti-HCV agents other than interferon/RBV and/or pegylated interferon (pegIFN)/RBV (including but not limited to telaprevir, boceprevir, sofosbuvir and simeprevir).
4. Confirmed presence of hepatocellular carcinoma indicated on imaging techniques such as CT scan or MRI within 3 months prior to Screening or on an ultrasound performed at Screening (a positive ultrasound result will be confirmed with CT scan or MRI).
5. Any current or past evidence of Child-Pugh C classification.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Cohen, MD, Study Director — AbbVie

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Started | 9 | 24 | 3
Completed | 9 | 22 | 2
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: GT1B: ombitasvir/paritaprevir/ritonavir 25/150/100 mg QD + dasabuvir 250 mg BID + RBV for 12 weeks in HCV GT1b-infected participants
- Total: Total of all reporting groups
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4 | Total
Number analyzed (Participants) | 9 | 24 | 3 | 36
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 7 | 20 | 2 | 29
  >= 65 years | 2 | 4 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 1 | 10
  Male | 7 | 17 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants With Sustained Virologic Response 12 Weeks Post-Treatment (SVR12) in Group 1 and in Group 2
Description: SVR12, defined as HCV RNA < lower limit of quantification (LLOQ) in the SVR12 window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. Flanking imputation: for participants with missing HCV RNA at a visit who have an undetectable HCV RNA or unquantifiable HCV RNA at the preceding visit and the succeeding visit, the missing value was imputed as undetectable or unquantifiable. For SVR analyses, if there was no value in the window after the flanking imputation but there was an HCV RNA value after the window, then it was imputed into the SVR window. After above imputations were applied, if there was still no value in the window but there was an HCV RNA value from a local laboratory present, then it was imputed into the SVR window. Otherwise, participants with missing data were counted as failures. The 95% confidence interval was calculated using the Wilson score method.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent to treat population: all participants who received at least 1 dose of study drug; participants missing data = non-responders. See imputation details in the outcome measure description.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B
Number analyzed (Participants) | 9 | 24
percentage of participants | 100 [70.1 to 100.0] | 95.8 [79.8 to 99.3]

2. Secondary Outcome: Percentage of Participants With SVR12 in Group 3
Description: SVR12, defined as HCV RNA < LLOQ in the SVR12 window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. Flanking imputation: for participants with missing HCV RNA at a visit, who have an undetectable HCV RNA or unquantifiable HCV RNA at the preceding visit and the succeeding visit, the missing value was imputed as undetectable or unquantifiable. For SVR analyses, if there was no value in the window after the flanking imputation but there was an HCV RNA value after the window, then it was imputed into the SVR window. After above imputations were applied, if there was still no value in the window but there was an HCV RNA value from a local laboratory present, then it was imputed into the SVR window. Otherwise, participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 3: GT4
Number analyzed (Participants) | 3
percentage of participants | 66.7

3. Secondary Outcome: Percentage of Participants With SVR12 Non-Response Due to Experiencing On-Treatment Virologic Failure
Description: On-treatment virologic failure was defined as: confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log˅10 IU/mL above nadir) at any time point during treatment; or HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks (≥ 36 days) of treatment. The 95% confidence interval was calculated using Wilson score method. SVR12 was defined as HCV RNA < LLOQ in the SVR12 window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window.
Time Frame: Up to 24 weeks during treatment
Population: Intent to treat population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 9 | 24 | 3
percentage of participants | 0 [0.0 to 29.9] | 0 [0.0 to 13.8] | 0 [NA to NA] — 95% confidence interval was not calculated for Group 3.

4. Secondary Outcome: Percentage of Participants With SVR12 Non-Response Due to Experiencing Relapse˅12
Description: Relapse˅12 was defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of active study drug (up to and including the SVR12 window) for a participant with HCV RNA < LLOQ at final treatment visit who completes treatment and has post-treatment HCV RNA data. Completion of treatment was defined as a study drug duration ≥ 77 days for participants assigned to 12 weeks of treatment or ≥ 154 days for participants assigned to 24 weeks of treatment. SVR12 was defined as HCV RNA < LLOQ in the SVR12 window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. The 95% confidence interval was calculated using the Wilson score method.
Time Frame: Up to 12 weeks after the last actual dose of study drug
Population: Intent to treat population: all participants who received at least 1 dose of study drug and who had an assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 7 | 19 | 2
percentage of participants | 0 [0.0 to 35.4] | 0 [0.0 to 16.8] | 0 [NA to NA] — 95% confidence interval was not calculated for Group 3.

5. Secondary Outcome: Percentage of Participants With Improvement From Baseline to Post-Treatment Week 12 in Hepatic Function Tests
Description: Improvement was defined as:
  * increase of more than 0.2 g/L from baseline to post-treatment Week 12 in albumin
  * decrease of more than 0.3 µmol/L from baseline to post-treatment Week 12 in bilirubin
  * decrease of more than 5 ng/mL from baseline to post-treatment Week 12 in alpha-fetoprotein
  * increase of more than 15*10^9/L from baseline to post-treatment Week 12 in platelet count
  * decrease of more than 0.2 from baseline to post-treatment Week 12 in international normalized ratio.
Time Frame: Up to post-treatment Week 12
Population: Intent to treat population: all participants who received at least 1 dose of study drug with values at both baseline and post-treatment Week 12 for the respective parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 9 | 22 | 2
percentage of participants
  Albumin | 77.8 | 77.3 | 50.0
  Bilirubin | 66.7 | 72.7 | 100
  Alpha-fetoprotein: number analyzed (Participants) | 9 | 0 | 0
  Alpha-fetoprotein | 33.3 |  |
  Platelet count: number analyzed (Participants) | 9 | 21 | 2
  Platelet count | 22.2 | 14.3 | 0
  International normalized ratio: number analyzed (Participants) | 9 | 21 | 2
  International normalized ratio | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Improvement From Baseline to Post-Treatment Week 12 in FibroTest
Description: The FibroTest score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis. Improvement was defined as a decrease of more than 0.2 from baseline to post-treatment Week 12.
Time Frame: Up to post-treatment Week 12
Population: Intent to treat population: all participants who received at least 1 dose of study drug with values at both baseline and post-treatment Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 9 | 22 | 2
percentage of participants | 0 | 9.1 | 50.0

7. Secondary Outcome: Percentage of Participants With Improvement From Baseline to Post-Treatment Week 12 in Chld-Pugh Score
Description: The The Child-Pugh score uses five clinical measures of liver disease (3 laboratory parameters and 2 clinical assessments) to measure severity of cirrhosis. Scores range from 5 to 15, with higher scores indicating more severity. Improvement was defined as a decrease of 1 or more from baseline to post-treatment Week 12.
Time Frame: Up to post-treatment Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 9 | 22 | 2
percentage of participants | 66.7 | 54.5 | 50.0

8. Secondary Outcome: Percentage of Participants With Improvement From Baseline to Post-Treatment Week 12 in Model for End-Stage Liver Disease (MELD) Score
Description: MELD is a scoring system for assessing the severity of chronic liver disease. Scores range from 6 to 40, with higher scores indicating more severity. Improvement was defined as a decrease of 1 or more from baseline to post-treatment Week 12.
Time Frame: Up to post-treatment Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Number analyzed (Participants) | 8 | 21 | 2
percentage of participants | 87.5 | 61.9 | 100

ADVERSE EVENTS:
Time Frame: Protocol-related treatment-emergent adverse events and treatment-emergent serious adverse events were collected from the first dose of study drug until post treatment Day 30; treatment was up to Week 12 for Group 1, and up to Week 24 for Groups 2 and 3.
Description: A protocol-related event is defined as any event with onset or worsening reported by a participant from the first dose of study drug until 30 days have elapsed following discontinuation of study drug administration. Events were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Group 1: GT1B | Group 2: GT1 Non-B | Group 3: GT4
Serious Adverse Events (participants affected / at risk) | 1/9 | 10/24 | 1/3
Other Adverse Events (participants affected / at risk) | 8/9 | 24/24 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: GT1B (N=9) | Group 2: GT1 Non-B (N=24) | Group 3: GT4 (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 1 | 1
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 2 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: GT1B (N=9) | Group 2: GT1 Non-B (N=24) | Group 3: GT4 (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 6 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 3 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 | 1
ASCITES (Gastrointestinal disorders) | 0 | 8 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 5 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 10 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 2 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 13 | 2
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 2 | 0
VOMITING (Gastrointestinal disorders) | 1 | 6 | 1
ASTHENIA (General disorders) | 0 | 4 | 1
CHILLS (General disorders) | 1 | 2 | 0
FATIGUE (General disorders) | 3 | 11 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 6 | 1
PYREXIA (General disorders) | 1 | 3 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 3 | 1
JAUNDICE (Hepatobiliary disorders) | 2 | 2 | 1
OCULAR ICTERUS (Hepatobiliary disorders) | 2 | 5 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 3 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 | 2 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 3 | 1
WEIGHT INCREASED (Investigations) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 5 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 7 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
DIZZINESS (Nervous system disorders) | 1 | 7 | 2
HEADACHE (Nervous system disorders) | 1 | 5 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 4 | 1
HYPERAESTHESIA (Nervous system disorders) | 0 | 0 | 1
HYPOTONIA (Nervous system disorders) | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 2 | 0
RADIAL NERVE PALSY (Nervous system disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
TREMOR (Nervous system disorders) | 1 | 3 | 0
ANXIETY (Psychiatric disorders) | 1 | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 1
INSOMNIA (Psychiatric disorders) | 0 | 6 | 2
IRRITABILITY (Psychiatric disorders) | 0 | 2 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 2
BREAST PAIN (Reproductive system and breast disorders) | 0 | 0 | 1
EJACULATION FAILURE (Reproductive system and breast disorders) | 0 | 0 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 7 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 7 | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.